CLINICAL TRIAL: NCT02904499
Title: Use of Public Health Surveillance Models in the French National Health System Database: A Tool for an Ongoing Monitoring of Adverse Drug Reaction? The Case of Dabigatran
Brief Title: Use of Public Health Surveillance Models in the French National Health System Database
Acronym: DABI-SURV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Principal Investigator, Laetitia HUIART, Methodologist, Centre Hospitalier Universitaire de la Réunion
Other Study IDs: 2012/CHU/01
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation; Anticoagulants; Pharmacoepidemiology
Keywords: Atrial Fibrillation; Anticoagulants; Pharmacoepidemiology
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- VKA: First Initiators of VKA for non-valvular atrial fibrilation
- Dabigatran: First Initiators of Dabigatran for non-valvular atrial fibrilation
  Interventions: Drug: Dabigatran

INTERVENTIONS:
Drug: Dabigatran
  Groups: Dabigatran

SUMMARY:
Public health surveillance models, previously used for the ongoing detection of occurrence of rare events, could be used to reinforce existing pharmacovigilance systems. These models have not been previously used for Adverse Drug Reaction (ADR) detection in medico-administrative databases. DABISURV research project focuses on a new anticoagulant therapy, dabigatran, launched recently on the French market for atrial fibrillation (AF). This drug is at high risk for severe ADR and requires thus careful pharmacovigilance monitoring.

Primary objective is to compare the results of ongoing surveillance models to detect hemorrhages or acute myocardial infarction (AMI) associated with dabigatran, with the results obtained from the analysis of a cohort of patients with AF under the same treatment.

DETAILED DESCRIPTION:
DABISURV study consists in an analyze of a cohort of patients with AF who have received at least one prescription Vitamin K Antagonists (VKA) - reference group - or of dabigatran in the French National Health Insurance System.

The uptake of dabigatran is followed for detecting hemorrhagic events or AMI associated with this molecule among first users.

The ability to detect quickly substantial ADR of new drugs is of critical importance to public health in order to facilitate timely public health response. If the public health surveillance models are found useful for this topic, then semi-automated procedures would be needed to detect ADR associated with new generation anticoagulants in medico-administrative databases. If the public health surveillance models are found not useful for the detection of ADR, the cohort study itself will provide essential data on the safety profile of dabigatran.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-valvular atrial fibrillation
* Patients receiving an first prescription of anticoagulants

Exclusion Criteria:

* Patients with valvular atrial fibrillation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of adult patients diagnosed with AF or atrial flutter and who received at least one prescription of VKA (warfarin /acenocoumarol /fluindion) or dabigatran between 2009 and 2014. As opposed to other countries, in France, warfarin is not the most prescribed VKA for AF.
Sampling Method: Probability Sample
Enrollment: 814446 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
results of ongoing surveillance models to detect hemorrhages or AMI (in frequency and proportion) associated with dabigatran or VKA for AF in a health database cohort of patients with AF treated by dabigatran or VKA | 36 months
  Propensity-matching is required for adequate comparison and multivariate regression

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Reunion Island, Saint-Denis, Reunion Island, France